CLINICAL TRIAL: NCT03383614
Title: A Phase 1, Single-Blind, Randomized, Placebo Controlled, Parallel-Group, Multiple-Dose-Escalation Study to Investigate Safety, Tolerability, and Pharmacokinetics of Emodepside (BAY 44-4400) After Oral Dosing in Healthy Male Subjects
Brief Title: Safety, Tolerability and PK of Multiple-ascending Doses of Emodepside
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Bayer (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNDI-EMO-02; 2017-003020-75 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2017-12-26 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Filariasis
MeSH Terms: conditions — Filariasis | interventions — Bay 44-4400

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort 1 (8 subjects) (Experimental): 6 subjects with LSF emodepside 5mg, OD 2 subjects with matching placebo
  Interventions: Drug: LSF emodepside (BAY 44-4400) or matching placebo
- cohort 2 (8 subjects) (Experimental): 6 subjects with LSF emodepside 10mg, OD 2 subjects with matching placebo
  Interventions: Drug: LSF emodepside (BAY 44-4400) or matching placebo
- cohort 3 (8 subjects) (Experimental): 6 subjects with LSF emodepside 10mg, BID 2 subjects with matching placebo
  Interventions: Drug: LSF emodepside (BAY 44-4400) or matching placebo

INTERVENTIONS:
Drug: LSF emodepside (BAY 44-4400) or matching placebo — Emodepside administered as an LSF oral solution (1mg/mL)

SUMMARY:
The study evaluates safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of emodepside, after administration as a Liquid Service Formulation (LSF), over 10 days, in healthy male caucasian subjects.

DETAILED DESCRIPTION:
There is an urgent need for a macrofilaricidal drug, killing or sterilizing permanently O. volvulus adult worms, which could be used in individual case management and, after appropriate testing, as an alternative drug to ivermectin in Mass Drug Administration (MDA) programs. Emodepside is a promising candidate to kill the adult and sexually mature O. volvulus as explained below. Emodepside was shown to be macrofilaricidal against a variety of filarial nematodes and is a registered drug for animal health, commercialized by Bayer AG under the name of Profender® (in combination with praziquantel) or Procox® (in combination with toltrazuril).

A first-in-human (FIH) double-blind, placebo-controlled study of single ascending doses of emodepside in healthy Caucasian men has been conducted and the preliminary results are favourable, supporting continuation of the Phase I development program. In the present repeat dose study, PK as well as safety and tolerability of the liquid service formulation of emodepside, given over 10 days, will be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Male, Caucasian volunteers, deemed healthy based on a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine.
2. 18 to 45 years of age.
3. Normal body weight (BMI; Quetelet index) in the range 18 to 30.1 kg/m2 at screening.
4. Blood pressure and heart rate in the supine position prior to randomisation must be within the ranges 90-140 mm Hg systolic, 60-90 mm Hg diastolic; heart rate 45-100 beats/min.
5. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial.
6. Willingness to give written consent to participate, after reading the information and consent form, and after having the opportunity to discuss the trial with the Investigator or his delegate.
7. Willingness to give written consent to have data entered into the Overvolunteering Prevention System.
8. Willingness to agree to the contraceptive requirements of the study from the first dose until 120 days after the last dose of study medication.

Exclusion Criteria:

1. Administration of a licensed or unlicensed medicinal product as part of another clinical trial within the 3 months before, or within 5 half-lives of, their first dose of study medication, whichever is longer, or is currently in the follow-up period for any clinical trial.
2. Clinically relevant abnormal medical history, concurrent medical condition, acute or chronic illness or history of chronic illness (such as diabetes mellitus or other abnormalities of glucose homeostasis) sufficient to invalidate the subject's participation in the trial or make it unnecessarily hazardous.
3. Past surgery (e.g., stomach bypass) or medical condition that might affect absorption of study drug taken orally.
4. Presence of abnormal physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the subject.
5. Loss of more than 400 mL of blood within 3 months before admission.
6. Clinically relevant history of vital organ disease or other disease of an organ or the central nervous system.
7. Current or previous medical or psychiatric disorder, condition or history of such (e.g., seizures) that, in the opinion of the Investigator or the Sponsor, would increase the risk associated with study participation, or impair the subject's ability to participate or complete this study.
8. Positive test for hepatitis B, hepatitis C or HIV.
9. Febrile illness within 1 week before the first dose of study medication.
10. History of severe allergy, non-allergic drug reactions, severe adverse reaction to any drug, or multiple drug allergies.
11. Subjects with hypersensitivity to any ingredient of the study medication, including the active ingredient, emodepside.
12. Presence or history of drug or alcohol abuse in the last 10 years, or intake of more than 21 units of alcohol weekly.
13. Regular daily consumption of more than one liter of xanthine-containing beverages.
14. Regular daily consumption of more than 5 cigarettes daily, or use more than 3 grams (1/8 ounce) of tobacco.
15. Use of a prescription medicine during the 28 days before the first dose of study medication or use of an over-the-counter medicine (with exception of acetaminophen [paracetamol]), during the 7 days before the first dose of study medication.
16. Use of dietary supplements or herbal remedies (such as St John's Wort) that are known to be inducers or inhibitors of CYP3A4, or other co-medications known to be relevant substrates of CYP3A4, during the 28 days before the first dose of study medication (see list in the Study Procedures Manual).
17. Use of dietary supplements or herbal remedies (such as St John's Wort) that are known to be strong inhibitors of P-gp, or other co-medications known to be relevant substrates of P-gp, during the 28 days before the first dose of study medication (see list in the Study Procedures Manual).
18. Relevant pathological abnormalities in the ECG at screening, such as a second or third-degree atrioventricular (AV) block or prolongation of the QRS complex over 120 msec or QTc-interval over 450 msec (corrected using Bazett's [QTcB] or Fridericia's [QTcF] formulae).
19. Evidence of drug abuse (via urine testing) at the screening assessment or admission to the ward.
20. Use of excluded therapies that may impact on the interpretation of study results in the opinion of the Investigator or Sponsor.
21. Objection by General Practitioner (GP) to subject entering trial.
22. History of residing for 6 or more continuous months, within the last 3 years, in regions with endemic parasitic infections as determined by the Investigator.
23. Possibility that subject will not cooperate with the requirements of the protocol.
24. No contact lenses wear within 1 month before dosing. Wearing contact lenses is not permitted during the study.
25. Any ocular disorder for which topical ocular therapy is currently or chronically prescribed, including inflammatory eye disease (dry eye allergic conjunctivitis [seasonal allergic conjunctivitis, vernal keratoconjunctivitis, atopic keratoconjunctivitis], uveitis and glaucoma).
26. Past history of ocular disease requiring ongoing treatment.
27. Past ocular surgery including laser or other refractive corneal surgery.
28. Evidence of eye irritation, visual difficulties, corneal opacity, ocular surface (corneal or conjunctival damage, with or without ocular symptoms).
29. Evidence of narrow anterior chamber angles causing increased risk of acute glaucoma.
30. Evidence of ocular media opacity including lens opacity/vitreous opacities.
31. Evidence of retinal or optic nerve pathology.
32. Evidence of pronounced colour blindness, as indicated by an Ishihara score of 9/13 or below.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only male subjects will be included
Enrollment: 24 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dennison, PhD MBChB, Principal Investigator — Hammersmith Medicines Research Limited
Locations (1):
- Hammersmith Medicines Research Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 healthy subjects were randomized and received study drug or matching placebo.
Groups:
- Cohort 1: 5mg EMODEPSIDE OD: 6 subjects with LSF emodepside 5mg, OD
  LSF emodepside (BAY 44-4400) oral solution (1mg/mL)
- Cohort 2: 10mg EMODEPSIDE OD: 6 subjects with LSF emodepside 10mg, OD
  LSF emodepside (BAY 44-4400) oral solution (1mg/mL)
- Cohort 3: 10mg EMODEPSIDE BID: 6 subjects with LSF emodepside 10mg, BID
  LSF emodepside (BAY 44-4400) oral solution (1mg/mL)
- Placebo Group: 6 subjects with matching placebo (2 subjects per dose group)
Period: Overall Study
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Started | 6 | 6 | 6 | 6
Completed | 6 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31.0 [19 to 41] | 33.3 [19 to 42] | 28.0 [20 to 43] | 32.7 [27 to 41] | 31.3 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 24
Height [Mean (Standard Deviation); unit: cm] | 179.3 (4.18) | 179.7 (4.59) | 181.8 (6.74) | 182.7 (8.80) | 180.9 (6.10)
Weight [Mean (Standard Deviation); unit: kg] | 72.18 (6.204) | 77.70 (17.570) | 75.23 (9.520) | 74.73 (8.999) | 74.96 (10.807)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.48 (2.520) | 23.88 (4.392) | 22.72 (2.111) | 22.33 (0.882) | 22.85 (2.664)
Smokers [Count of Participants; unit: Participants] — Includes only those subjects who smoked.
  Participants | 2 | 1 | 1 | 0 | 4
Weekly alcohol consumption (units) [Mean (Standard Deviation); unit: units/week] — Population: Includes only those subjects who drank alcohol-containing beverages.
  units/week
    number analyzed (Participants) | 3 | 3 | 4 | 5 | 15
    (all) | 8.3 (3.79) | 3.3 (2.31) | 7.0 (3.46) | 5.8 (2.17) | 6.1 (3.11)
Xanthine [Mean (Standard Deviation); unit: mL/day] — Population: Includes only those subjects who drank xanthine-containing beverages.
  mL/day
    number analyzed (Participants) | 6 | 4 | 3 | 6 | 19
    (all) | 441.7 (245.80) | 562.5 (239.36) | 283.3 (104.08) | 300.0 (122.47) | 397.4 (209.15)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Adverse Events
Description: Death, serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs).
Time Frame: up to 120 days
Population: Adverse events were determined in the Safety population. Adverse events were monitored from Screening (Day -28 and until Day -3) to Follow-up (up to Day 120 ±2 days).
  AE=adverse event; OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  AEs | 5 | 6 | 6 | 4
  TEAEs | 5 | 6 | 6 | 4
  Drug-related TEAEs | 2 | 1 | 3 | 1
  SAEs | 1 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0
  Withdrawals from the study owing to a TEAE | 0 | 0 | 0 | 0

2. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Adverse Event Severity
Description: Number of subjects with a TEAE, by highest level of severity.
Time Frame: Up to 120 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Mild | 2 | 3 | 4 | 3
  Moderate | 2 | 3 | 2 | 1
  Severe | 1 | 0 | 0 | 0

3. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Vital Signs Findings
Description: Vital signs included heart rate, systolic and diastolic blood pressure and temperature.
Time Frame: up to 120 days
Population: Vital signs were measured pre-dose on Day -1, at regular time points until Follow-up (Day 30), and at each long-term follow-up visit.
  OD=once daily; BID=twice daily; HR=heart rate; BP=blood pressure.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Clinically significant change in HR | 0 | 0 | 0 | 0
  Clinically significant change in systolic BP | 0 | 0 | 0 | 0
  Clinically significant change in diastolic BP | 0 | 0 | 0 | 0
  Clinically significant change in temperature | 0 | 0 | 0 | 0

4. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With 12-lead Electrocardiogram Findings
Description: The following variables were recorded in 12-lead ECGs: ventricular rate, PR interval, QRS interval, QTcB and QTcF interval.
Time Frame: up to 30 days
Population: Twelve-lead ECG assessments were made predose on Day -1 and at regular timepoints until Follow-up (Day 30).
  ECG=electrocardiogram; OD=once daily; BID=twice daily; PR=PR interval.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Clinically significant changes in ventricular rate | 0 | 0 | 0 | 0
  Clinically significant changes in PR interval | 0 | 0 | 0 | 0
  Clinically significant changes in QRS interval | 0 | 0 | 0 | 0
  Clinically significant changes in QTcB interval | 0 | 0 | 0 | 0

5. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Clinical Laboratory Tests Findings
Description: Clinical laboratory parameters included clinical chemistry, hematology, coagulation and urinalysis.
Time Frame: up to 120 days
Population: Clinical laboratory parameters were measured pre-dose on Day -1, at regular time points until Follow-up (Day 30), and at each long-term follow-up visit.
  OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Clinically significant clinical chemistry changes | 0 | 0 | 1 | 0
  Clinically significant hematology changes | 0 | 0 | 0 | 0
  Clinically significant coagulation changes | 0 | 0 | 0 | 0
  Clinically significant urinalysis changes | 0 | 0 | 0 | 0

6. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Ophthalmology Assessment Findings
Description: Ophthalmological examinations at Screening Visit 2 and Day 10 were done at a specialist eye hospital by a Consultant Ophthalmologist, or their assistant. Examinations included: ocular symptoms and history, autorefraction, best correct visual acuity, colour vision, Amsler grid, ocular alignment and motility, confrontation visual field, slit-lamp, measurement of intraocular pressure and an optical coherence tomography test.
Time Frame: up to 10 days
Population: Ophthalmological assessments were performed at the second screening visit after all other eligibility criteria had been met and on Day 10.
  OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Clinically significant ocular symptoms | 3 | 0 | 3 | 1
  Clinically significant Amsler grid assessment | 1 | 0 | 0 | 0

7. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Physical Examination Findings
Description: Abnormal or clinically significant physical examination findings during the study or reported as an adverse event.
Time Frame: up to 120 days
Population: Physical and neurological examinations were measured pre-dose on Day -1, at regular time points until Follow-up (Day 30), and at each long-term follow-up visit. Results are reported for subjects experiencing abnormal result/AE, as opposed to individual events.
  OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Abnormal physical examination | 2 | 1 | 2 | 0
  Physical examination reported as an AE | 2 | 1 | 1 | 0

8. Primary Outcome: Safety and Tolerability of Emodepside After Multiple Doses as Measured by Number of Participants With Neurological Examination Findings
Description: Abnormal or clinically significant neurological examination findings during the study or reported as an adverse event.
Time Frame: up to 120 days
Population: Neurological examinations were measured pre-dose on Day -1, at regular time points until Follow-up (Day 30), and at each long-term follow-up visit.
  OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Abnormal neurological examination | 2 | 1 | 1 | 1
  Neurological examination reported as an AE | 1 | 1 | 1 | 1

9. Secondary Outcome: Geometric Mean Emodepside Plasma Pharmacokinetic Concentration-Time Data During the Repeated Dosing Period
Description: Summary of geometric mean emodepside plasma pharmacokinetic concentration-time data (ng/mL) during the repeated dosing period (Days 0-9) in healthy men.
  Subjects in the 10 mg emodepside BID dosing group had twice-daily doses on Days 0-8 and a single dose on the morning of Day 9. Therefore, the Day 9, 24 h post-dose value was not comparable to the previous value in that dosing group.
Time Frame: From Day 1, pre-dose to Day 9, 24 hours post-dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1: Emodepside 5 mg OD: Emodepside (BAY 44-4400) 5 mg orally, once daily in fasted state.
- Cohort 2: Emodepside 10 mg OD: Emodepside (BAY 44-4400) 10 mg orally, once daily in fasted state.
- Cohort 3: Emodepside 10 mg BID: Emodepside (BAY 44-4400) 10 mg orally, twice a day (morning and evening) in fasted state.
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day 1, pre-dose | 8.77 (35.8) | 15.78 (42.9) | 45.94 (35.1)
  Day 2, pre-dose | 15.24 (31.1) | 28.80 (40.0) | 64.62 (38.5)
  Day 3, pre-dose | 21.22 (35.0) | 39.08 (45.6) | 84.65 (37.7)
  Day 4, pre-dose | 24.81 (37.4) | 47.38 (42.2) | 98.01 (32.0)
  Day 5, pre-dose | 31.46 (36.3) | 60.07 (42.9) | 120.98 (31.1)
  Day 6, pre-dose | 36.68 (36.7) | 70.88 (39.6) | 137.60 (35.2)
  Day 7, pre-dose | 40.57 (31.4) | 83.31 (43.0) | 149.41 (33.3)
  Day 8, pre-dose | 46.91 (36.8) | 91.63 (42.4) | 179.90 (35.3)
  Day 9, pre-dose | 49.73 (35.1) | 97.11 (44.0) | 184.94 (37.1)
  Day 9, 24 hour post-dose | 51.76 (36.6) | 108.17 (49.1) | 176.10 (39.8)

10. Secondary Outcome: The AUClast of Emodepside in Plasma
Description: Summary of AUClast of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUClast: the area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration.
  PK=pharmacokinetic. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUClast in plasma after the last dose (Day 9)
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 19359 (29.9) | 40655 (43.5) | 59554 (29.1)

11. Secondary Outcome: The AUClast/D of Emodepside in Plasma
Description: Summary of AUClast/D of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUClast/D: the area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration corrected for dose.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUClast /D in plasma after the last dose (Day 9)
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL/mg | 3872 (29.9) | 4065 (43.5) | 5955 (29.1)

12. Secondary Outcome: The AUClast,Norm of Emodepside in Plasma
Description: Summary of AUClast,norm of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUClast,norm: the area under the concentration-time curve from time zero (pre-dose) to the time of last quantifiable concentration corrected by dose and body weight.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUClast,norm in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/(mg*kg)
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
(h*ng/mL)/(mg*kg) | 53.9 (33.1) | 52.9 (69.5) | 79.1 (40.6)

13. Secondary Outcome: The AUC12 of Emodepside in Plasma
Description: Summary of AUC12 of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUC12: the area under the concentration-time curve from time zero (pre-dose) to 12h.
  Note: AUC12 was calculated only in Cohort 3. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC12 in plasma after the first (Day 0) and last (Day 9) dose
Population: BID=twice daily.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6
h*ng/mL
  Day 0 | 742 (29.4)
  Day 9 | 2810 (35.0)

14. Secondary Outcome: The AUC12/D of Emodepside in Plasma
Description: Summary of AUC12/D of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUC12/D: the area under the concentration-time curve from time zero (pre-dose) to 12h, corrected for dose.
  Note: AUC12/D was collected only in Cohort 3. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC12/D in plasma after the first (Day 0) and last (Day 9) dose
Population: BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6
h*ng/mL/mg
  Day 0 | 74.2 (29.4)
  Day 9 | 281 (35.0)

15. Secondary Outcome: The AUC12,Norm of Emodepside in Plasma
Description: Summary of AUC12,norm of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  AUC12,norm: the area under the concentration-time curve from time zero (pre-dose) to 12 h corrected by dose and body weight.
  Note: AUC12,norm was calculated only in Cohort 3. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC12,norm in plasma after the first (Day 0) and last (Day 9) dose
Population: BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/(mg*kg)
Arm/Group | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6
(h*ng/mL)/(mg*kg)
  Day 0 | 0.985 (39.2)
  Day 9 | 3.73 (46.6)

16. Secondary Outcome: The AUC24 of Emodepside in Plasma
Description: Summary of AUC24 of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  AUC24: the area under the concentration-time curve from time zero (pre-dose) to 24 h.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC24 in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL
  Day 0 | 574 (19.7) | 1135 (32.7) | 1428 (26.5)
  Day 9 | 1689 (31.3) | 3487 (44.2) | 4897 (35.8)

17. Secondary Outcome: The AUC24/D of Emodepside in Plasma
Description: Summary of AUC24/D of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  AUC24/D: the area under the concentration-time curve from time zero (pre-dose) to 24h corrected for dose.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC24/D in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL/mg
  Day 0 | 115 (19.7) | 113 (32.7) | 71.4 (26.5)
  Day 9 | 338 (31.3) | 349 (44.2) | 490 (35.8)

18. Secondary Outcome: The AUC24,Norm of Emodepside in Plasma
Description: Summary of AUC24,norm of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120h (Day 14) after the morning dose.
  AUC24,norm: the area under the concentration-time curve from time zero (pre-dose) to 24h corrected by dose and body weight.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: AUC24,norm in plasma at Day 0 and Day 9
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (h*ng/mL)/(mg*kg)
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
(h*ng/mL)/(mg*kg)
  Day 0 | 1.60 (21.5) | 1.48 (56.7) | 0.948 (36.5)
  Day 9 | 4.70 (34.1) | 4.54 (69.7) | 6.50 (47.7)

19. Secondary Outcome: The Cmax of Emodepside in Plasma
Description: Summary of Cmax of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  Cmax: the observed maximum plasma concentration measured in a subject after dosing identified by inspection of the drug concentration vs. time data.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: Cmax in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Day 0 | 93.8 (17.8) | 186 (21.3) | 160 (20.4)
  Day 9 | 149 (17.9) | 287 (39.7) | 349 (27.1)

20. Secondary Outcome: The Cmax/D of Emodepside in Plasma
Description: Summary of Cmax/D of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  Cmax/D: the observed maximum plasma concentration measured in a subject after dosing identified by inspection of the drug concentration vs. time data, corrected for dose.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: Cmax/D in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
ng/mL/mg
  Day 0 | 18.8 (17.8) | 18.6 (21.3) | 16.0 (20.4)
  Day 9 | 29.9 (17.9) | 28.7 (39.7) | 34.9 (27.1)

21. Secondary Outcome: The Cmax,Norm of Emodepside in Plasma
Description: Summary of Cmax,norm of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  Cmax,norm: the observed maximum plasma concentration measured in a subject after dosing identified by inspection of the drug concentration vs. time data, corrected for dose and body weight.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: Cmax,norm in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)*(mg*kg)
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
(ng/mL)*(mg*kg)
  Day 0 | 0.261 (18.4) | 0.242 (42.8) | 0.212 (28.7)
  Day 9 | 0.416 (20.6) | 0.374 (65.4) | 0.464 (38.2)

22. Secondary Outcome: The Ctrough of Emodepside in Plasma
Description: Summary of Ctrough (log-transformed) of emodepside after last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  Ctrough: trough plasma concentration (measured concentration at the end of a dosing interval on Day 9 [taken directly before next administration]) obtained directly from the concentration-time data.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: Ctrough in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 49.7 (36.8) | 97.1 (50.8) | 185 (39.5)

23. Secondary Outcome: The Tmax of Emodepside in Plasma
Description: Summary of tmax of emodepside after the first (Day 0) and last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose. Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  tmax: the time at which Cmax was apparent, identified by inspection of the drug concentration vs. time data.
Time Frame: tmax in plasma after the first (Day 0) and last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Hours
  Day 0 | 1.00 [1.00 to 1.07] | 1.25 [1.00 to 2.00] | 1.00 [1.00 to 1.58]
  Day 9 | 1.00 [1.00 to 1.50] | 1.25 [1.00 to 2.00] | 1.50 [1.03 to 2.50]

24. Secondary Outcome: The t1/2 of Emodepside in Plasma
Description: Summary of t1/2 of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  t1/2: terminal half-life. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: t1/2 in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Hours | 419 (42.6) | 450 (30.6) | 508 (56.9)

25. Secondary Outcome: The t1/2,(0-24) of Emodepside in Plasma
Description: Summary of t1/2,(0-24) of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  t1/2,(0-24): half-life calculated from the terminal slope of the log concentration-time (0-24h) curve.
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: t1/2,(0-24) in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Hours | 26.9 (52.4) | 18.4 (30.0) | 33.2 (55.0)

26. Secondary Outcome: The λz of Emodepside in Plasma
Description: Summary of λz of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  λz: terminal rate constant. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: λz in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
1/h | 0.00166 (42.6) | 0.00154 (30.6) | 0.00137 (56.9)

27. Secondary Outcome: The CLss/F of Emodepside in Plasma
Description: Summary of CLss/F of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  CLss/F: apparent total clearance from plasma on Day 9. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: CLss/F in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
L/h | 2.96 (31.3) | 2.87 (44.2) | 3.56 (35.0)

28. Secondary Outcome: The Vz/F of Emodepside in Plasma
Description: Summary of Vz/F of emodepside after the last (Day 9) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 9 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 15, 24, 36 (Day 10), 48 (Day 11), 72 (Day 12), 96 (Day 13) and 120 h (Day 14) after the morning dose.
  Vz/F: apparent volume of distribution on Day 9. The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: Vz/F in plasma after the last (Day 9) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre(s)
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
litre(s) | 1788 (74.2) | 1861 (68.5) | 2607 (102.1)

29. Secondary Outcome: The MRTlast of Emodepside in Plasma
Description: Summary of MRTlast of emodepside after the first (Day 0) dose for 10-day oral treatment courses in healthy men: PK parameter population.
  Data on Day 0 was collected at the following time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 15 h after the morning dose.
  MRTlast: mean residence time from time zero (pre-dose) to the time of last quantifiable concentration (measurable up to 24h after dosing on Day 0).
  The geometric coefficient of variation is the between-subject coefficient of variation (%CVb).
Time Frame: MRTlast in plasma after the first (Day 0) dose
Population: OD=once daily; BID=twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Hours | 7.28 (10.7) | 7.00 (11.0) | 10.8 (2.8)

30. Secondary Outcome: The Rac(AUC12) of Emodepside in Plasma
Description: Summary of emodepside plasma Rac(AUC12) after 10 days' repeated doses of 10 mg emodepside (Day 9): PK parameter population.
  Rac(AUC12): accumulation ratio calculated from AUC12, where AUC12 is the area under the concentration-time curve from time zero (pre-dose) to 12h.
  Note: measure of dispersion is 'percentage coefficient of variation' (the between-subject coefficient of variation [%CVb]).
  Note: Rac(AUC12) was calculated only in Cohort 3.
Time Frame: Rac(AUC12) after 10 days' repeated doses of 10 mg emodepside (Day 9)
Population: BID=twice daily.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6
Ratio | 3.83 (15.5)

31. Secondary Outcome: The Rac(AUC24) of Emodepside in Plasma
Description: Summary of emodepside plasma Rac(AUC24) after 10 days' repeated doses of 10 mg emodepside (Day 9): PK parameter population.
  Rac(AUC24): accumulation ratio calculated from AUC24, where AUC24 is the area under the concentration-time curve from time zero (pre-dose) to 24h.
  Note: measure of dispersion is 'percentage coefficient of variation' (the between-subject coefficient of variation [%CVb]).
Time Frame: Rac(AUC24) after 10 days' repeated doses of 10 mg emodepside (Day 9)
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 2.97 (16.1) | 3.09 (11.3) | 3.47 (17.1)

32. Secondary Outcome: The Rac(Cmax) of Emodepside in Plasma
Description: Summary of emodepside plasma Rac(Cmax) after 10 days' repeated doses of 10 mg emodepside (Day 9): PK parameter population.
  Rac(Cmax): accumulation ratio calculated from Cmax, where Cmax is the observed maximum plasma concentration measured in a subject after dosing identified by inspection of the drug concentration vs. time data.
  Note: measure of dispersion is 'percentage coefficient of variation' (the between-subject coefficient of variation [%CVb]).
Time Frame: Rac(Cmax) after 10 days' repeated doses of 10 mg emodepside (Day 9)
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1: Emodepside 5 mg OD | Cohort 2: Emodepside 10 mg OD | Cohort 3: Emodepside 10 mg BID
Number analyzed (Participants) | 6 | 6 | 6
Ratio | 1.61 (16.5) | 1.58 (24.1) | 2.21 (17.4)

33. Secondary Outcome: Mean Glucose Concentration at Day -1
Description: Mean glucose concentrations (mmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day -1.
Time Frame: Mean glucose at Day -1 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  -24 h | 4.72 (0.286) | 4.68 (0.349) | 4.80 (0.245) | 4.77 (0.468)
  -23 h: number analyzed (Participants) | 5 | 6 | 6 | 6
  -23 h | 4.90 (0.308) | 4.85 (0.259) | 4.85 (0.281) | 4.92 (0.313)
  -22 h | 4.77 (0.378) | 4.72 (0.371) | 4.72 (0.279) | 4.82 (0.360)
  -20 h | 4.63 (0.388) | 4.57 (0.207) | 4.55 (0.207) | 4.73 (0.480)
  -12 h | 5.17 (0.712) | 5.55 (0.451) | 5.52 (0.556) | 5.48 (0.806)

34. Secondary Outcome: Mean Glucose Concentration at Day 0
Description: Mean glucose concentrations (mmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 0.
  Baseline=predose on Day 0.
Time Frame: Mean glucose after repeated once or twice daily dosing for up to 10 days
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  Predose (Baseline): number analyzed (Participants) | 5 | 6 | 6 | 6
  Predose (Baseline) | 4.96 (0.321) | 4.85 (0.409) | 4.85 (0.351) | 4.85 (0.288)
  1 h | 5.07 (0.367) | 5.57 (0.816) | 5.42 (0.445) | 4.78 (0.214)
  2 h | 5.05 (0.327) | 5.28 (0.508) | 5.27 (0.472) | 4.70 (0.310)
  4 h | 4.73 (0.378) | 4.75 (0.274) | 4.82 (0.279) | 4.70 (0.276)
  12 h: number analyzed (Participants) | 5 | 6 | 6 | 6
  12 h | 5.68 (0.268) | 6.22 (0.343) | 5.57 (0.554) | 6.27 (0.761)
  24 h | 5.07 (0.314) | 4.88 (0.264) | 4.87 (0.273) | 4.97 (0.288)

35. Secondary Outcome: Mean Glucose Concentration at Day 9
Description: Mean glucose concentrations (mmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 9.
Time Frame: Mean glucose at Day 9 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  Predose | 4.52 (0.306) | 4.95 (0.362) | 4.97 (0.314) | 4.67 (0.234)
  1 h: number analyzed (Participants) | 6 | 5 | 6 | 6
  1 h | 5.10 (0.352) | 5.98 (1.972) | 5.65 (0.771) | 4.80 (0.219)
  2 h: number analyzed (Participants) | 6 | 6 | 6 | 5
  2 h | 5.03 (0.250) | 5.72 (1.543) | 5.57 (0.761) | 4.74 (0.329)
  4 h: number analyzed (Participants) | 6 | 5 | 6 | 6
  4 h | 4.60 (0.363) | 4.62 (0.377) | 5.08 (0.662) | 4.70 (0.374)
  12 h: number analyzed (Participants) | 6 | 5 | 6 | 6
  12 h | 5.58 (0.319) | 6.00 (0.745) | 7.03 (1.111) | 6.02 (0.615)
  24 h | 4.92 (0.264) | 5.10 (0.490) | 5.17 (0.273) | 4.82 (0.160)
  48 h | 5.02 (0.194) | 5.07 (0.532) | 5.10 (0.390) | 4.90 (0.379)
  72 h | 4.87 (0.350) | 5.13 (0.589) | 5.03 (0.308) | 5.03 (0.280)
  96 h | 4.80 (0.276) | 5.10 (0.540) | 4.85 (0.315) | 4.87 (0.320)
  120 h | 5.00 (0.352) | 4.98 (0.458) | 5.05 (0.288) | 4.90 (0.352)

36. Secondary Outcome: Mean Glucose Concentration at Day 30
Description: Mean glucose concentrations (mmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 30.
Time Frame: Mean glucose at Day 30 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L | 4.83 (0.288) | 5.23 (0.993) | 4.97 (0.234) | 4.53 (0.350)

37. Secondary Outcome: Mean Insulin Concentration at Day -1
Description: Mean insulin concentration (pmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day -1.
Time Frame: Mean insulin concentration at Day-1 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  -24 h | 29.0 (8.60) | 25.8 (8.11) | 33.2 (17.90) | 32.3 (12.31)
  -23 h | 25.8 (3.87) | 26.2 (7.73) | 28.0 (11.33) | 26.5 (8.92)
  -22 h | 24.0 (6.69) | 25.7 (8.91) | 28.3 (14.50) | 33.0 (5.73)
  -20 h | 22.7 (6.02) | 22.7 (7.97) | 24.3 (9.18) | 24.5 (12.76)
  -12 h | 129.5 (54.14) | 157.0 (81.51) | 204.7 (78.37) | 136.5 (64.30)

38. Secondary Outcome: Mean Insulin Concentration at Day 0
Description: Mean insulin concentration (pmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 0.
  Baseline=predose on Day 0.
Time Frame: Mean insulin concentration at Day 0 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  Predose (Baseline) | 27.8 (15.41) | 29.3 (5.09) | 32.2 (14.34) | 30.5 (12.55)
  1 h | 25.0 (3.79) | 23.2 (10.85) | 29.2 (14.86) | 33.0 (9.10)
  2 h | 24.3 (5.20) | 25.3 (9.99) | 36.3 (20.39) | 31.2 (12.89)
  4 h | 21.7 (5.01) | 21.7 (5.39) | 27.7 (11.69) | 20.2 (6.85)
  12 h | 127.2 (67.59) | 203.2 (83.22) | 175.3 (64.59) | 195.0 (88.03)
  24 h | 36.7 (15.49) | 41.2 (14.51) | 30.3 (11.43) | 35.2 (16.59)

39. Secondary Outcome: Mean Insulin Concentration at Day 9
Description: Mean insulin concentration (pmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 9.
Time Frame: Mean insulin concentration at Day 9 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  Predose | 31.5 (8.62) | 32.7 (15.02) | 29.2 (10.19) | 31.3 (9.83)
  1 h: number analyzed (Participants) | 6 | 5 | 6 | 6
  1 h | 29.2 (9.66) | 24.4 (15.39) | 22.2 (8.89) | 27.8 (9.77)
  2 h: number analyzed (Participants) | 6 | 6 | 6 | 5
  2 h | 27.7 (4.84) | 31.2 (10.53) | 30.2 (13.91) | 29.8 (10.26)
  4 h: number analyzed (Participants) | 6 | 5 | 6 | 6
  4 h | 23.0 (7.35) | 28.4 (13.24) | 19.5 (9.12) | 21.8 (6.37)
  12 h | 147.2 (77.58) | 143.0 (113.7) | 215.8 (128.1) | 215.7 (151.8)
  24 h | 34.5 (11.88) | 36.5 (12.24) | 32.7 (17.44) | 36.3 (13.03)
  48 h | 36.2 (5.60) | 44.8 (17.89) | 36.3 (13.59) | 38.2 (19.17)
  72 h | 48.3 (23.53) | 40.7 (13.88) | 39.8 (15.61) | 38.7 (14.42)
  96 h | 37.8 (10.42) | 39.3 (12.31) | 37.2 (17.66) | 30.0 (11.63)
  120 h | 39.0 (8.63) | 42.3 (17.92) | 36.0 (15.24) | 33.2 (21.68)

40. Secondary Outcome: Mean Insulin Concentration at Day 30
Description: Mean insulin concentration (pmol/L) after repeated once or twice daily dosing with up to 10 mg emodepside or placebo at Day 30.
Time Frame: Mean insulin concentration at Day 30 after repeated once or twice daily dosing
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L | 29.2 (12.50) | 60.3 (90.19) | 24.3 (9.79) | 29.2 (20.21)

41. Secondary Outcome: Mean Serum Glucose Concentration at Day -2
Description: Oral glucose tolerance test: mean serum glucose concentration at Day -2, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum glucose concentration at Day -2, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  0 h (Baseline) | 4.72 (0.319) | 4.92 (0.256) | 4.97 (0.294) | 4.78 (0.133)
  1 h | 8.78 (1.659) | 7.03 (0.301) | 7.00 (0.867) | 6.48 (1.450)
  2 h | 5.98 (1.512) | 5.05 (0.589) | 5.48 (0.608) | 4.95 (0.965)
  4 h | 4.57 (0.979) | 3.95 (0.622) | 4.22 (0.371) | 4.53 (0.294)

42. Secondary Outcome: Mean Serum Glucose Concentration at Day 1
Description: Oral glucose tolerance test: mean serum glucose concentration at Day 1, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum glucose concentration at Day 1, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  Predose (Baseline) | 5.07 (0.314) | 4.88 (0.264) | 4.87 (0.273) | 4.97 (0.228)
  1 h | 10.10 (1.170) | 12.37 (2.826) | 12.03 (0.989) | 7.58 (2.242)
  2 h | 6.17 (1.600) | 7.95 (1.653) | 9.25 (2.740) | 5.88 (1.174)
  4 h | 3.95 (0.339) | 3.65 (0.362) | 4.02 (0.204) | 4.15 (0.575)

43. Secondary Outcome: Mean Serum Glucose Concentration at Day 8
Description: Oral glucose tolerance test: mean serum glucose concentration at Day 8, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum glucose concentration at Day 8, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmol/L
  Predose (Baseline) | 4.87 (0.314) | 5.10 (0.533) | 4.90 (0.303) | 4.83 (0.258)
  1 h | 10.02 (1.857) | 11.75 (4.574) | 11.27 (2.738) | 7.77 (1.679)
  2 h | 7.05 (1.533) | 8.98 (4.311) | 8.97 (2.837) | 5.52 (0.783)
  4 h | 3.93 (0.965) | 4.12 (0.933) | 4.52 (0.806) | 4.13 (0.197)

44. Secondary Outcome: Mean Serum Glucose Concentration at Day 120
Description: Oral glucose tolerance test: mean serum glucose concentration at Day 120, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day. Note: At Day 120, serum glucose concentration was only measured in Cohort 3 (10 mg BID)
Time Frame: Mean serum glucose concentration at Day 120, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 3: 10mg EMODEPSIDE BID
Number analyzed (Participants) | 6
mmol/L
  0 h (Baseline) | 4.93 (0.294)
  1 h: number analyzed (Participants) | 5
  1 h | 8.12 (2.542)
  2 h: number analyzed (Participants) | 5
  2 h | 6.08 (0.540)
  4 h: number analyzed (Participants) | 5
  4 h | 4.26 (0.305)

45. Secondary Outcome: Mean Serum Insulin Concentration at Day -2
Description: Oral glucose tolerance test: mean serum insulin concentration at Day -2, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum insulin concentration at Day -2, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  0 h (Baseline) | 24.5 (13.81) | 25.7 (8.55) | 27.0 (14.00) | 29.0 (14.68)
  1 h | 334.8 (207.66) | 305.3 (65.59) | 306.7 (180.00) | 338.3 (189.61)
  2 h | 174.7 (206.08) | 103.7 (32.38) | 136.0 (70.52) | 186.8 (83.55)
  4 h | 44.3 (72.56) | 17.2 (6.11) | 20.8 (7.44) | 21.8 (9.33)

46. Secondary Outcome: Mean Serum Insulin Concentration at Day 1
Description: Oral glucose tolerance test: mean serum insulin concentration at Day 1, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum insulin concentration at Day 1, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  Predose (Baseline) | 36.7 (15.49) | 41.2 (14.51) | 30.3 (11.43) | 35.2 (16.59)
  1 h | 312.2 (153.67) | 288.8 (171.44) | 332.2 (228.84) | 606.7 (157.35)
  2 h | 268.5 (107.14) | 377.3 (224.73) | 336.2 (165.71) | 238.0 (165.06)
  4 h | 28.8 (22.35) | 30.8 (12.35) | 35.7 (4.59) | 33.8 (19.56)

47. Secondary Outcome: Mean Serum Insulin Concentration at Day 8
Description: Oral glucose tolerance test: mean serum insulin concentration at Day 8, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day.
Time Frame: Mean serum insulin concentration at Day 8, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
pmol/L
  Predose (Baseline) | 32.5 (9.85) | 39.3 (22.59) | 34.5 (15.83) | 33.8 (12.94)
  1 h | 302.5 (145.61) | 286.8 (179.53) | 225.3 (148.93) | 690.5 (342.10)
  2 h | 337.0 (110.23) | 225.7 (101.02) | 229.8 (79.00) | 238.3 (92.34)
  4 h | 63.0 (86.69) | 63.3 (83.32) | 36.8 (21.17) | 21.7 (19.97)

48. Secondary Outcome: Mean Serum Insulin Concentration at Day 120
Description: Oral glucose tolerance test: mean serum insulin concentration at Day 120, before and up to 4 hours after intake of a high-glucose solution, in subjects receiving repeated doses of emodepside or placebo for 10 days (Days 0-9).
  Baseline=pre-glucose intake on each respective day. Note: At Day 120, serum glucose concentration was only measured in Cohort 3 (10 mg BID)
Time Frame: Mean serum insulin concentration at Day 120, before and up to 4 hours after intake of a high-glucose solution
Population: OD=once daily; BID=twice daily.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Cohort 3: 10mg EMODEPSIDE BID
Number analyzed (Participants) | 6
pmol/L
  0 h (Baseline) | 28.0 (13.74)
  1 h: number analyzed (Participants) | 5
  1 h | 417.8 (379.72)
  2 h: number analyzed (Participants) | 5
  2 h | 152.8 (114.92)
  4 h: number analyzed (Participants) | 5
  4 h | 18.8 (11.39)

49. Other Pre Specified Outcome: Drug-related Adverse Events
Description: Subjects presenting drug-related treatment-emergent adverse events listed by preferred term.
  Note: subjects with ≥1 adverse event are counted only once per preferred term.
Time Frame: Drug-related AEs were reported throughout the study
Population: OD=once daily; BID=twice daily.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Visual impairment | 2 | 1 | 3 | 1
  Euphoric mood | 1 | 1 | 0 | 0
  Nervousness | 1 | 0 | 0 | 0
  Dizziness | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from Screening (Day -28 and until Day -3) to Follow-up (up to Day 120 ±2 days).
Arm/Group | Cohort 1: 5mg EMODEPSIDE OD | Cohort 2: 10mg EMODEPSIDE OD | Cohort 3: 10mg EMODEPSIDE BID | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 6/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 5mg EMODEPSIDE OD (N=6) | Cohort 2: 10mg EMODEPSIDE OD (N=6) | Cohort 3: 10mg EMODEPSIDE BID (N=6) | Placebo Group (N=6)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The fistula was downgraded by the investigator to a nonserious AE on 05 NOV 2018; after final database lock. That decision was based on the fact that the subject was hospitalised because of the AE of anal abscess, and not the fistula.
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 5mg EMODEPSIDE OD (N=6) | Cohort 2: 10mg EMODEPSIDE OD (N=6) | Cohort 3: 10mg EMODEPSIDE BID (N=6) | Placebo Group (N=6)
Sebaceous cyst excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E antibody positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (4)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 2 (3) | 1 (2) | 3 (3) | 1 (1)
Vision blurred (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT03383614/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT03383614/SAP_001.pdf